CLINICAL TRIAL: NCT02603146
Title: Strategy to Prevent the Onset of Clinically-Apparent Rheumatoid Arthritis
Acronym: StopRA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment was closed before reaching the target. In the 1st interim analysis after enrollment closure, the follow up & treatment of active participants were stopped early due to evidence of futility.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DAIT ARA08; NIAID CRMS ID#: 20681 (Other: DAIT NIAID)
Record Dates: First submitted 2015-11-10; First posted 2015-11-11 (Estimated); Results first posted 2023-11-21 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Healthy Participants; Rheumatoid Arthritis (RA) Prevention
Keywords: RA prevention; hydroxychloroquine (HCQ); anti-CCP3
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydroxychloroquine Group (Experimental): Subjects randomized to hydroxychloroquine (HCQ). Subjects will receive 200-400 mg of HCQ (1-2 pills), based upon ideal body weight (IBW), taken daily for 12 months.
  Interventions: Drug: Hydroxychloroquine
- Placebo Group (Placebo Comparator): Subjects randomized to placebo HCQ. Subjects will receive 200 - 400 mg of HCQ placebo (1-2 pills), based upon IBW, taken daily for 12 months.
  Interventions: Drug: HCQ Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — As described. Dosing will be based upon Screening IBW.
  Other Names: HCQ; Plaquenil
  Arms: Hydroxychloroquine Group
Drug: HCQ Placebo — As described. Dosing will be based upon Screening IBW.
  Other Names: Placebo
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to determine if hydroxychloroquine (HCQ) is safe and effective for the prevention of future onset of rheumatoid arthritis (RA) in individuals who have elevations of an autoantibody, anti-cyclic citrullinated peptide (anti-CCP3).

The following recruitment strategies will be employed towards identifying healthy subjects with elevated anti-cyclic citrullinated peptide (anti-CCP3) levels:

-Pre-screening:

* first degree relatives of patients with rheumatoid arthritis (RA);
* subjects at health-fairs; and
* identification of subjects with elevated anti-CCP3 levels in the absence of inflammatory arthritis in rheumatology clinics.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) affects an estimated 1% of the population. RA is a disease where the immune system attacks the joints, leading to joint inflammation and damage that is felt by someone with RA as joint pain, stiffness and swelling.

Recent studies have shown that there are markers in the blood called 'autoantibodies' that precede the onset of joint symptoms of RA. Antibodies are commonly made in the blood to fight infections. Sometimes, these antibodies attack one's own body. These are called autoantibodies.

Certain autoantibodies are specific for certain diseases. The autoantibody known as anti-CCP3 is specific for RA and can predict the development of RA in the future, especially if the level of anti-CCP3 is high. The investigators of this study believe that individuals with elevations of anti-CCP3 ≥2 times the normal value have approximately a 50% chance of developing RA within 3 years.

Hydroxychloroquine (HCQ) is already used successfully and safely in the treatment of malaria, lupus and RA. The objective of this study is to determine whether treatment with HCQ in individuals with elevations of anti-CCP3 without joint inflammation may help prevent the future onset of RA. This will involve a 12-month course of HCQ in the prevention of the development of clinically apparent RA at 36 months in individuals at high-risk for future RA due to high titer elevations of anti-CCP3. This study will recruit for individuals without a history or clinical findings of inflammatory arthritis. Eligible subjects will be randomized in a 1:1 ratio to HCQ versus HCQ placebo.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria are eligible for enrollment into the study:

* Able and willing to give written informed consent and comply with requirements of the study;
* Age ≥18 years-old at the Screening Visit; and
* Elevation of autoantibody anti-cyclic citrullinated peptide-3 (anti-CCP3) defined by result of anti-CCP3 ≥40 units, at Screening.

Exclusion Criteria:

Subjects who meet any of the following criteria are ineligible to participate in the study:

-A medical history of inflammatory arthritis (IA) of any type and/or rheumatic disease and immunologic disease(s) that may be associated with IA . These diseases include but are not limited to:

* rheumatoid arthritis (RA);
* systemic lupus erythematosus (SLE);
* seronegative spondyloarthropathies;
* inflammatory bowel disease;
* Sjögren's syndrome;
* polymyalgia rheumatic; or
* vasculitis.

Note: Crystalline arthropathies are not exclusionary.

* A medical history of:

  * congestive heart failure or functional status of New York Heart Association (NYHA) Class III or higher at the Screening Visit;
  * cardiomyopathy or significant cardiac conduction disorders;
  * chronic liver disease;
  * psoriasis (due to potential for increased risk for flare of skin disease);
  * porphyria;
  * and/or serologic evidence during Screening Visit of chronic infections including, but not limited to, human immunodeficiency virus (HIV), hepatitis B (HBV), hepatitis C (HCV);

    ---Exception: hepatitis C antibody positive subjects are eligible with documentation of:
    * receipt of HCV treatment AND
    * a negative hepatitis C viral load test post-treatment.
  * malignancy within the last 5 years, except for treated basal or squamous cell carcinoma, treated cervical dysplasia, or treated in situ cervical cancer Grade I; or
  * alcohol or substance abuse within 1 year of treatment randomization.
* Prior or current systemic treatment with disease modifying anti-rheumatic agents, immunomodulatory agents, or glucocorticoids for IA, other rheumatic diseases, or other immunologic diseases;
* Tetracycline class antibiotic use for autoimmune conditions, taken within 12 months prior to Screening;
* Systemic corticosteroid use for non-IA conditions taken 28 days prior to Screening;
* More than 3 local corticosteroid injections, including but not limited to intra-articular, epidural, and intrabursal injections, during the 3 months prior to randomization;
* A history of a chronic condition that, in the opinion of the investigator, is highly likely to require therapy with systemic corticosteroids (oral or intravenous) within the study period, including but not limited to severe asthma and severe crystalline arthropathy;
* Women who are pregnant, breastfeeding or desire to become pregnant and/or breast feed within the duration of the 12-month treatment phase of the study;
* Women of childbearing potential who are not using or who do not agree to use adequate birth control measures (for example, total abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, surgical sterilization, Depo-Provera, or hormonal implants) during the treatment phase of the study;
* An ideal or actual body weight ≤ 24.4 kg (e.g., ≤53 lbs) at Screening Visit;
* Any of the following laboratory abnormalities at the Screening Visit:

  * Serum Creatinine Clearance < 50ml/min (as calculated by the Cockcroft-Gault formula: Creatinine clearance (CrCl)= (140-age) X (Weight in kg) X (0.85 if female) / (72 X Creatinine));
  * Alanine Aminotransferase (ALT) > 2 times the upper limit of normal (ULN);
  * Aspartate Aminotransferase (AST) > 2x the upper limit of normal (ULN);
  * Total white blood count (WBC) < 3.0 x 10^9/L;
  * Platelet count ≤ 150 x10^9/L;
  * Hemoglobin < 11.5g/dL;
  * Absolute Neutrophil Count (ANC) < 2.0 x 10^9/L;
* Evidence of significant retinal disease upon eye examination during the screening period that in the opinion of the examiner would make identification of potential future retinal toxicity from HCQ difficult to evaluate:

  -- Retinal exam results may be applied to evaluations of subject eligibility for up to 6 months after the initial retinal exam.
* When, in the opinion of the study physician, the subject is not a good study candidate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Deane, MD, PhD, Study Chair — University of Colorado School of Medicine; Michael Holers, MD, Study Chair — University of Colorado School of Medicine; Christopher Striebich, MD, PhD, Study Chair — University of Colorado School of Medicine
Locations (14):
- United States (14):
  - University of Alabama at Birmingham School of Medicine: Division of Clinical Immunology & Rheumatology, Birmingham, Alabama
  - Cedars Sinai Medical Center: Division of Rheumatology, Los Angeles, California
  - UCLA Medical Center: Division of Rheumatology, Los Angeles, California
  - University of California San Francisco, San Francisco General Hospital, San Francisco, California
  - University of Colorado School of Medicine: Division of Rheumatology, Aurora, Colorado
  - Emory Clinic at 1365 Clifton Road: Emory University School of Medicine, Atlanta, Georgia
  - Brigham & Women's Hospital: Department of Medicine, Rheumatology, Immunology, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center: Rheumatology, Worcester, Massachusetts
  - University of Michigan Health System: Department of Internal Medicine, Division of Rheumatology, Ann Arbor, Michigan
  - Mayo Clinic, Division of Rheumatology, Rochester, Minnesota
  - University of Nebraska Medical Center: Division of Rheumatology, Omaha, Nebraska
  - Northwell Health, Great Neck, New York
  - Oklahoma Medical Research Foundation: Arthritis and Clinical Immunology Research Program, Oklahoma City, Oklahoma
  - University of Texas Southwestern Medical Center, Division of Rheumatic Diseases, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data in ImmPort, a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts, upon completion of the trial.
Time Frame: After completion of the study.
Access Criteria: When posted, the IPD will be available to the public.
URL: http://www.immport.org/

REFERENCES:
- [Derived] Deane KD, Striebich CC, Feser ML, O'Dell JR, James JA, Sparks JA, Davis JM, Graf J, McMahon MA, Solow EB, Forbess L, Tiliakos A, Schiopu E, Danila MI, Horowitz DL, Kay J, Strickland CD, Guthridge JM, Arriens C, Grossman JM, Demoruelle MK, Bemis EA, Frazer-Abel A, Fleischer CL, Fox DA, Mikuls TR, Greenleaf M, York K, Walker S, Keyes-Elstein L, Byron M, Fedler J, Goldmuntz EA, Holers VM. A phase 2 trial of hydroxychloroquine in individuals at risk for rheumatoid arthritis. Arthritis Rheumatol. 2025 Aug 29. doi: 10.1002/art.43366. Online ahead of print. PMID 40884017
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty study sites were activated in the United States, beginning in March 2016. A total of 252 participants were screened from April 2016 to October 2021 at 15 sites. 144 participants were randomized.
Groups:
- Hydroxychloroquine: Participants self-administered 1-2 200 mg HCQ pills per day, based on ideal body weight at screening, from the Baseline visit to Week 52.
- Placebo: Participants self-administered 1-2 placebo pills per day, based on ideal body weight at screening, from the Baseline visit to Week 52.
Period: Overall Study
Arm/Group | Hydroxychloroquine | Placebo
Started | 71 | 73
Completed | 40 | 39
Not Completed | 31 | 34
Not completed — Lost to Follow-up | 5 | 6
Not completed — Withdrawal by Subject | 8 | 10
Not completed — Withdrawn by Investigator or NIAID | 15 | 18
Not completed — Participant moved | 2 | 0
Not completed — Participant could not complete the Month 36 visit due to COVID-19 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat population includes all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxychloroquine | Placebo | Total
Number analyzed (Participants) | 71 | 73 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 61 | 120
  >=65 years | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (12.31) | 49.3 (14.39) | 50.5 (13.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 58 | 115
  Male | 14 | 15 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 8 | 23
  Not Hispanic or Latino | 55 | 64 | 119
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 6 | 14
  White | 53 | 55 | 108
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 71 | 73 | 144
Anti-Cyclic Citrullinated Peptide-3 (Anti-CCP3) [Mean (Standard Deviation); unit: units] — Anti-CCP3 is a laboratory test for the presence of antibodies to citrullinated protein antigens (ACPAs) in serum. ACPA positivity assists with the classification/diagnosis of Rheumatoid Arthritis (RA) of a patient with Inflammatory Arthritis (IA). In addition, determining autoantibody positivity helps with the prediction of RA disease severity. Anti-CCP3 positivity at any level, and in particular anti-CCP3 levels of ≥2 times the normal cut-off level (or ≥ 40 units) are highly predictive of future RA development. A value above 40 units was required to enter the study.
  units | 173.2 (86.01) | 147.4 (86.42) | 160.1 (86.89)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed Clinically-Apparent Rheumatoid Arthritis (CL - RA) From Treatment Initiation to Month 36 By Treatment Arm
Description: Clinically-Apparent RA is defined by the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) Classification Criteria as either: 1.) a score of ≥ 6 defining "definite RA" or 2.) a joint examination consistent with Inflammatory Arthritis (IA) with ≥ 1 erosion confirmed by x-ray imaging of the hands, wrists, and feet.
Time Frame: Baseline to Month 36
Population: The modified-intent-to-treat population includes all randomized participants who received at least one dose of assigned study drug and met entry criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 69 | 73
Participants | 20 | 24
Statistical Analysis 1: Comparison: Hydroxychloroquine; Test type: Other; Cumulative Probability = 0.336, 95% CI 2-sided [0.213 to 0.459] — Using Kaplan-Meier product-limit method (and Greenwood's formula for confidence interval), estimated the cumulative probability of development of CL-RA by Month 36 for HCQ
Statistical Analysis 2: Comparison: Placebo; Test type: Other; Cumulative Probability = 0.394, 95% CI 2-sided [0.268 to 0.519] — Using Kaplan-Meier product-limit method (and Greenwood's formula for confidence interval), estimated the cumulative probability of development of CL-RA by Month 36 for Placebo
Statistical Analysis 3: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority — The analysis is based on the KM estimated risk of CL- RA at 36 months, where risk = (1-KM estimated probability of "survival"). Survival for this analysis is defined as absence of CL-RA. Estimated risks were derived from a Kaplan-Meier curve using censored time-to-event data to account for attrition under the assumption of non-informative censoring; p = 0.522, Chi-squared — The test statistic is a Wald-type chi-square statistic derived by dividing the difference of the logit-transformed KM survival estimates for each arm by the associated variance derived using the delta-method [Klein, et. al. 2007]; Risk Difference (RD) = -0.058, 95% CI 2-sided [-0.336 to 0.220] — Risk difference for HCQ - Placebo

2. Secondary Outcome: Number of Participants Who Developed Clinically-Apparent Rheumatoid Arthritis (CL-RA) From Treatment Initiation to Month 12 By Treatment Arm
Description: Clinically-Apparent RA is defined by the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) Classification Criteria as either: 1.) a score of ≥ 6 defining "definite RA" or 2.) a joint examination consistent with IA with ≥ 1 erosion confirmed by x-ray imaging of the hands, wrists, and feet.
Time Frame: Baseline to Month 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 69 | 73
Participants | 11 | 13
Statistical Analysis 1: Comparison: Hydroxychloroquine; Test type: Other; Cumulative Probability = 0.165, 95% CI 2-sided [0.076 to 0.225] — Using Kaplan-Meier product-limit method (and Greenwood's formula for confidence interval), estimated the cumulative probability of development of CL-RA by Month 12 for HCQ
Statistical Analysis 2: Comparison: Placebo; Test type: Other; Cumulative Probability = 0.194, 95% CI 2-sided [0.099 to 0.289] — Using Kaplan-Meier product-limit method (and Greenwood's formula for confidence interval), estimated the cumulative probability of development of CL-RA by Month 12 for Placebo
Statistical Analysis 3: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority — The analysis is based on the KM estimated risk of CL- RA at 12 months, where risk = (1-KM estimated probability of "survival"). Survival for this analysis is defined as absence of CL-RA. Estimated risks were derived from a Kaplan-Meier curve using censored time-to-event data to account for attrition under the assumption of non-informative censoring; p = 0.668, Chi-squared — [p-value comment as in outcome 1, analysis 3]; Risk Difference (RD) = -0.029, 95% CI 2-sided [-0.188 to 0.131] — Risk difference for HCQ - Placebo

3. Secondary Outcome: Number of Participants Who Developed Inflammatory Arthritis (IA) From Treatment Initiation to Month 12.
Description: IA is defined as the development of at least one swollen joint consistent with rheumatoid arthritis-like (RA-like) synovitis. The joint exams conducted by a physician at each clinic visit were used to identify the presence of swollen joints due to IA.
Time Frame: Baseline to Month 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 69 | 73
Participants | 12 | 13
Statistical Analysis 1: Comparison: Hydroxychloroquine; Test type: Other; Cumulative Probability = 0.180, 95% CI 2-sided [0.088 to 0.273] — Using Kaplan-Meier product-limit method (and Greenwood's formula for confidence interval), estimated the cumulative probability of development of IA by Month 12 for HCQ
Statistical Analysis 2: Comparison: Placebo; Test type: Other; Cumulative Probability = 0.194, 95% CI 2-sided [0.099 to 0.289] — Using Kaplan-Meier product-limit method (and Greenwood's formula for confidence interval), estimated the cumulative probability of development of IA by Month 12 for Placebo
Statistical Analysis 3: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority — The analysis is based on the KM estimated risk of IA at 12 months, where risk = (1-KM estimated probability of "survival"). Survival for this analysis is defined as absence of IA. Estimated risks were derived from a Kaplan-Meier curve using censored time-to-event data to account for attrition under the assumption of non-informative censoring; p = 0.840, Chi-squared — [p-value comment as in outcome 1, analysis 3]; Risk Difference (RD) = -0.014, 95% CI 2-sided [-0.177 to 0.150] — Risk difference for HCQ - Placebo

4. Secondary Outcome: Time to Development of Clinically-Apparent Rheumatoid Arthritis (CL - RA) By Treatment Arm
Description: Mean Time from treatment initiation until development of CL-RA. CL- RA is defined by the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) Classification Criteria as either: 1.) a score of ≥ 6 defining "definite RA" or 2.) a joint examination consistent with IA with ≥ 1 erosion confirmed by x-ray imaging of the hands, wrists, and feet.
Time Frame: Baseline to Month 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 69 | 73
months | 29.02 [25.84 to 32.21] | 28.49 [25.40 to 31.58]
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; p = 0.652, Log Rank

5. Secondary Outcome: Number of Participants Who Developed Inflammatory Arthritis (IA) From Treatment Initiation to Month 36
Description: as for outcome 3
Time Frame: Baseline to Month 36
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 69 | 73
Participants | 21 | 27
Statistical Analysis 1: Comparison: Hydroxychloroquine; Test type: Other; Cumulative Probability = 0.356, 95% CI 2-sided [0.230 to 0.482] — Using Kaplan-Meier product-limit method (and Greenwood's formula for confidence interval), estimated the cumulative probability of development of IA by Month 36 for HCQ
Statistical Analysis 2: Comparison: Placebo; Test type: Other; Cumulative Probability = 0.425, 95% CI 2-sided [0.298 to 0.551] — Using Kaplan-Meier product-limit method (and Greenwood's formula for confidence interval), estimated the cumulative probability of development of IA by Month 36 for Placebo
Statistical Analysis 3: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority — The analysis is based on the KM estimated risk of IA at 36 months, where risk = (1-KM estimated probability of "survival"). Survival for this analysis is defined as absence of IA. Estimated risks were derived from a Kaplan-Meier curve using censored time-to-event data to account for attrition under the assumption of non-informative censoring; p = 0.452, Chi-squared — [p-value comment as in outcome 1, analysis 3]; Risk Difference (RD) = -0.069, 95% CI 2-sided [-0.363 to 0.226] — Risk difference for HCQ - Placebo

6. Secondary Outcome: Number of Participant Self-Reported Painful Joints By Treatment Arm
Description: The Participant Self-Reported Joint Symptoms assessment was used by participants to indicate which joints were painful on the day of the visit or in the past week. The Participant Self-Reported Joint Symptoms assessment contained a diagram of the body joints which participants used to mark their painful joints.
Time Frame: At Week 52 and Month 36/End of Study
Population: Participants in the modified-intent-to-treat population, including all randomized participants who received at least one dose of assigned study drug and met entry criteria, and who have available data at the time point.
Measure: Median (Full Range); unit: joints
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 69 | 73
joints
  Week 52: number analyzed (Participants) | 53 | 57
  Week 52 | 1.0 [0 to 23] | 1.0 [0 to 38]
  Month 36: number analyzed (Participants) | 38 | 39
  Month 36 | 1.0 [0 to 13] | 2.0 [0 to 36]
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; p = 0.928, Wilcoxon (Mann-Whitney) — Week 52 results
Statistical Analysis 2: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; p = 0.076, Wilcoxon (Mann-Whitney) — Month 36 results

7. Secondary Outcome: Number of Participant Self-Reported Stiff Joints By Treatment Arm
Description: The Participant Self-Reported Joint Symptoms assessment was used by participants to indicate which joints were stiff on the day of the visit or in the past week. The Participant Self-Reported Joint Symptoms assessment contained a diagram of the body joints which participants used to mark their stiff joints.
Time Frame: At Week 52 and Month 36/End of Study
Population: as for outcome 6
Measure: Median (Full Range); unit: Joints
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 69 | 73
Joints
  Week 52: number analyzed (Participants) | 53 | 57
  Week 52 | 1.0 [0 to 32] | 1.0 [0 to 42]
  Month 36: number analyzed (Participants) | 38 | 39
  Month 36 | 0.0 [0 to 32] | 1.0 [0 to 20]
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; p = 0.781, Wilcoxon (Mann-Whitney) — Week 52 results
Statistical Analysis 2: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; p = 0.457, Wilcoxon (Mann-Whitney) — Month 36 results

8. Secondary Outcome: Number of Participant Self-Reported Swollen Joints By Treatment Arm
Description: The Participant Self-Reported Joint Symptoms assessment was used by participants to indicate which joints were swollen on the day of the visit or in the past week. The Participant Self-Reported Joint Symptoms assessment contained a diagram of the body joints which participants used to mark their swollen joints.
Time Frame: At Week 52 and Month 36/End of Study
Population: The modified-intent-to-treat population includes all randomized participants who received at least one dose of assigned study drug and met entry criteria, and who have available data at the time point.
Measure: Median (Full Range); unit: Joints
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 69 | 73
Joints
  Week 52: number analyzed (Participants) | 53 | 57
  Week 52 | 0.0 [0 to 8] | 0.0 [0 to 23]
  Month 36: number analyzed (Participants) | 38 | 39
  Month 36 | 0.0 [0 to 3] | 0.0 [0 to 24]
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; p = 0.576, Wilcoxon (Mann-Whitney) — Week 52 results
Statistical Analysis 2: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; p = 0.323, Wilcoxon (Mann-Whitney) — Month 36 results

9. Secondary Outcome: Number of Participant Self-Reported Painful Joints in the Hands, Wrists and Feet By Treatment Arm
Description: as for outcome 6
Time Frame: At Week 52 and Month 36/End of Study
Population: as for outcome 8
Measure: Median (Full Range); unit: Joints
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 69 | 73
Joints
  Week 52: number analyzed (Participants) | 53 | 57
  Week 52 | 0.0 [0 to 21] | 0.0 [0 to 32]
  Month 36: number analyzed (Participants) | 38 | 39
  Month 36 | 0.0 [0 to 11] | 0.0 [0 to 30]
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; p = 0.865, Wilcoxon (Mann-Whitney) — Week 52 results
Statistical Analysis 2: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; p = 0.179, Wilcoxon (Mann-Whitney) — Month 36 results

10. Secondary Outcome: Number of Participant Self-Reported Stiff Joints in the Hands, Wrists and Feet By Treatment Arm
Description: as for outcome 7
Time Frame: At Week 52 and Month 36/End of Study
Population: as for outcome 8
Measure: Median (Full Range); unit: Joints
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 69 | 73
Joints
  Week 52 results: number analyzed (Participants) | 53 | 57
  Week 52 results | 0.0 [0 to 22] | 0.0 [0 to 32]
  Month 36 results: number analyzed (Participants) | 38 | 39
  Month 36 results | 0.0 [0 to 22] | 12 [0 to 20]
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; p = 0.634, Wilcoxon (Mann-Whitney) — Week 52 results
Statistical Analysis 2: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; p = 0.574, Wilcoxon (Mann-Whitney) — Month 36 results

11. Secondary Outcome: Number of Participant Self-Reported Swollen Joints in the Hands, Wrists and Feet By Treatment Arm
Description: as for outcome 8
Time Frame: At Week 52 and Month 36/End of Study
Population: as for outcome 8
Measure: Median (Full Range); unit: Joints
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 69 | 73
Joints
  Week 52: number analyzed (Participants) | 53 | 57
  Week 52 | 0.0 [0 to 8] | 0.0 [0 to 21]
  Month 36: number analyzed (Participants) | 38 | 39
  Month 36 | 0.0 [0 to 3] | 0.0 [0 to 22]
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; p = 0.724, Wilcoxon (Mann-Whitney) — Week 52 results
Statistical Analysis 2: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; p = 0.149, Wilcoxon (Mann-Whitney) — Month 36 results

12. Secondary Outcome: Level of Anti-Cyclic Citrullinated Peptide-3 (Anti-CCP3) By Treatment Arm
Description: Anti-CCP3 is a laboratory test for the presence of antibodies to citrullinated protein antigens (ACPAs) in serum. ACPA positivity assists with the classification/diagnosis of Rheumatoid Arthritis (RA) of a patient with Inflammatory Arthritis (IA). In addition, determining autoantibody positivity helps with the prediction of RA disease severity. Anti-CCP3 positivity at any level, and in particular anti-CCP3 levels of ≥2 times the normal cut-off level (or ≥ 40 units) are highly predictive of future RA development.
Time Frame: Baseline, Week 52 (End of Treatment), Month 36/End of Study
Population: as for outcome 8
Measure: Median (Full Range); unit: units
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 69 | 73
units
  Baseline: number analyzed (Participants) | 69 | 72
  Baseline | 184.20 [24.3 to 261.7] | 125.55 [28.4 to 261.7]
  Week 52: number analyzed (Participants) | 44 | 50
  Week 52 | 105.65 [19.6 to 261.7] | 94.4 [17.9 to 261.7]
  Month 36: number analyzed (Participants) | 28 | 29
  Month 36 | 154.75 [15.2 to 261.7] | 85.20 [9.0 to 261.7]

13. Secondary Outcome: Level of Immunoglobulin M - Rheumatoid Factor (IgM-RF) By Treatment Arm
Description: IgM-RF is a laboratory test for the presence of antibodies to RF in serum. IgM-RF positivity assists with the classification/diagnosis of Rheumatoid Arthritis (RA) of a patient with Inflammatory Arthritis (IA). In addition, determining autoantibody positivity helps with the prediction of RA disease severity. Higher levels of antibodies (e.g. >2-3 times the normal cut-off values) have greater specificity for RA disease.
Time Frame: Baseline, Week 52 (End of Treatment), Month 36/End of Study
Population: as for outcome 8
Measure: Median (Full Range); unit: U/mL
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 69 | 73
U/mL
  Baseline: number analyzed (Participants) | 69 | 72
  Baseline | 13.100 [0.25 to 104.75] | 5.350 [0.14 to 104.75]
  Week 52: number analyzed (Participants) | 44 | 50
  Week 52 | 3.600 [0.25 to 104.75] | 2.025 [0.25 to 104.75]
  Month 36: number analyzed (Participants) | 28 | 29
  Month 36 | 5.730 [0.25 to 104.75] | 0.250 [0.25 to 104.75]

14. Secondary Outcome: Level of High-Sensitivity C-Reactive Protein (hsCRP) Treatment Arm
Description: HsCRP is used to detect systemic inflammation in the body, assists with the classification/diagnosis of Rheumatoid Arthritis (RA), and elevations of hsCRP in patients with RA have been associated with poor disease outcomes.
Time Frame: Baseline, Week 52 (End of Treatment), Month 36/End of Study
Population: as for outcome 8
Measure: Median (Full Range); unit: mg/L
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 69 | 73
mg/L
  Baseline: number analyzed (Participants) | 69 | 71
  Baseline | 2.030 [0.21 to 40.40] | 3.043 [0.13 to 43.70]
  Week 52: number analyzed (Participants) | 48 | 53
  Week 52 | 2.300 [0.20 to 56.30] | 1.430 [0.21 to 55.70]
  Month 36: number analyzed (Participants) | 34 | 35
  Month 36 | 2.075 [0.20 to 22.75] | 1.645 [0.27 to 29.50]

15. Secondary Outcome: Percent of Participants Experiencing Grade 3 or Higher Adverse Events (AEs)
Description: Adverse Events (AEs) grading will be defined by the National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events (CTCAE), version 4.0. The number of AEs will be identified by monitoring participant-reported AEs, vital signs, medical history, physical exams and blood safety tests.
Time Frame: Non-serious AEs were collected from treatment initiation through month 18. Serious AEs were collected from screening through month 36.
Population: The safety population includes all participants for whom study treatment was initiated.
Measure: Number; unit: Percent of Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 69 | 73
Percent of Participants | 14.1 | 12.3
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; p = 0.809, Fisher Exact

ADVERSE EVENTS:
Time Frame: Grade 2 or higher treatment-emergent adverse events were collected from the time of administration of the first dose of study drug (HCQ/placebo) until Month 18 or until 30 days after the participant prematurely withdrew (without withdrawing consent) or was withdrawn from the study, whichever occurred first. Serious adverse events were collected from the time of administration of the first dose of study drug until Month 36.
Arm/Group | Hydroxychloroquine | Placebo
All-Cause Mortality (participants affected / at risk) | 1/71 | 0/73
Serious Adverse Events (participants affected / at risk) | 5/71 | 5/73
Other Adverse Events (participants affected / at risk) | 25/71 | 31/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (N=71) | Placebo (N=73)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Desmoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (N=71) | Placebo (N=73)
Sinusitis (Infections and infestations) | 1 (1) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (5)
Urinary tract infection (Infections and infestations) | 5 (6) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 16 (16) | 19 (19)
Hypertension (Vascular disorders) | 7 (7) | 6 (6)

LIMITATIONS AND CAVEATS:
Enrollment closed at 144 randomized participants before reaching the target of 200 due to slow participant accrual. The decision was supported by a revised power analysis suggesting sufficient power for the study with reduced numbers assuming a clinically-relevant difference in RA rates between arms (50% risk for placebo & 25% risk for HCQ). In the 1st interim analysis after enrollment closure, the follow up & treatment of the active participants were stopped early due to evidence of futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT02603146/Prot_002.pdf
  • Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/46/NCT02603146/SAP_003.pdf